CLINICAL TRIAL: NCT04102917
Title: The Catholic Imaging and Functional Research Cohort (C-iFR)
Brief Title: Diagnostic Performance and Prognostic Ability of the QFR
Status: Completed | Type: Observational
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: National Research Foundation of Korea (Other); Seoul Saint Mary's Hospital (Unknown); Incheon Saint Mary's Hospital (Unknown); Seoul Saint Paul's Hospital (Unknown); Uijeongbu Saint Mary's Hospital (Unknown)
Responsible Party: Principal Investigator, Kiyuk Chang, Prof., Seoul St. Mary's Hospital
Other Study IDs: XC18REDI0035
Record Dates: First submitted 2019-09-15; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Ischemic Heart Disease
Keywords: QFR; quantitative flow ratio
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- QFR group: 915 patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, acute myocardial infarction with non-culprit stenosis who underwent FFR measurement and were able to analyze QFR.
  Interventions: Diagnostic Test: QFR assessment

INTERVENTIONS:
Diagnostic Test: QFR assessment — The quantitative flow ratio (QFR) is a novel angiography-based method for noninvasive functional assessment of intermediate coronary lesions.

SUMMARY:
1. The primary technical endpoint was the diagnostic performance of the QFR against the FFR.
2. The primary clinical endpoint was target vessel failure (TVF) between two groups distributed by a QFR cut-off value of 0.8

DETAILED DESCRIPTION:
The quantitative flow ratio (QFR) is a novel angiography-based tool used to assess functional ischemia caused by coronary stenosis. Computation of the fractional flow reserve (FFR) from coronary angiography is based on 3D reconstruction and fluid dynamics algorithms using a modified frame count; therefore, we do not need to induce hyperemia or perform invasive procedures with a pressure wire to measure it. During the past few years, the diagnostic accuracy of the QFR was investigated and showed favorable outcomes. However, data for patients with acute coronary syndrome are lacking. In addition, no data are available for the performance of the QFR in predicting clinical outcomes. We aim to evaluate the diagnostic performance of the QFR versus the FFR and their predictive abilities for clinical outcome in a real-world all-comer population.

The Catholic imaging and Functional Research (C-iFR) Cohort was designed to evaluate the diagnostic performance and clinical outcome predictive ability of the QFR in consecutive patients undergoing CAG and the FFR at 4 major cardiac centers in Korea from January 2012 to May 2018. All hospitals (Seoul St. Mary's Hospital, Seoul; St. Paul's Hospital, Seoul; Incheon St. Mary's Hospital, Incheon; Uijeongbu St. Mary's Hospital, Uijeongbu) perform a high volume of percutaneous coronary intervention (PCI) procedures, with more than 800 PCI procedures performed per year. This QFR registry includes demographic characteristics, clinical information, laboratory data, QFR findings, and FFR findings, with clinical outcome data collected over 4 years (a median of 2 years)

ELIGIBILITY:
Inclusion Criteria:

* subject ≥18 years
* Patients suspected with ischemic heart disease
* All-comer patients with SA, UA and AMI whose CAG results showed intermediate stenosis (50-70%) indicative of physiologic lesions
* Patients whose target vessels were able to analyze QFR

Exclusion Criteria: Patients with insufficient CAG data due to reasons below

* CAG data uploading error
* 2 projection angles <25 degrees apart
* only 1 projection angle image exists
* images with suboptimal contrast filling
* images with too much panning or too much magnification
* containing an ostial lesion of the left main coronary artery or right coronary artery
* anatomical vessel problems including severe overlap, severe tortuosity, foreshortening, diffuse lesions, additional far distal lesion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 915 patients with suspected ischemic heart disease including stable angina, or acute coronary syndrome including unstable angina, acute myocardial infarction with non-culprit stenotic lesion who underwent FFR measurement and were able to analyze QFR
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy, sensitivity, specificity, negative predictive value, positive predictive value of QFR | follow up of 4 years (anticipated median duration : 2 years)
  the diagnostic accuracy, sensitivity, specificity, negative predictive value, positive predictive value of the QFR≤0.80 for identifying an FFR≤0.8 as the reference standard
Target vessel failure | follow up of 4 years (anticipated median duration : 2 years)
  target vessel failure (TVF) between two groups distributed by a QFR cut-off value of 0.8

SECONDARY OUTCOMES:
Diagnostic accuracy, sensitivity, specificity, negative predictive value, positive predictive value of QFR in subgroups with a borderline FFR (≥0.75, ≤0.85) | follow up of 4 years (anticipated median duration : 2 years)
  the sensitivity, specificity, negative predictive value, positive predictive value of the QFR≤0.80 for identifying an FFR≤0.8 as the reference standard in subgroups with a borderline FFR (≥0.75, ≤0.85)
Diagnostic accuracy, sensitivity, specificity, negative predictive value, positive predictive value of QFR in subgroups with complicated coronary lesions | follow up of 4 years (anticipated median duration : 2 years)
  the sensitivity, specificity, negative predictive value, positive predictive value of the QFR≤0.80 for identifying an FFR≤0.8 as the reference standard in subgroups with complicated coronary lesions, such as bifurcation lesions, a large intraluminal plaque volume, a low mean flow rate, a long lesion length, calcification, tandem lesions, and a previous history of coronary intervention
All-cause death, cardiac death, nonfatal myocardial infarction, TLR and stroke | follow up of 4 years (anticipated median duration : 2 years)
  all-cause death, cardiac death, nonfatal myocardial infarction, TLR and stroke between two groups distributed by a QFR cut-off value of 0.80

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, MD, PhD, Principal Investigator — Seoul Saint Mary's Hospital
Locations (1):
- Seoul Saint Mary's Hospital, Seoul, Seochogu, South Korea

IPD SHARING:
Plan to Share IPD: No